CLINICAL TRIAL: NCT02502422
Title: Prediction of Optimal Laryngeal Mask Airway Cuff Volume From Parameters of Physical Examination of Head and Neck
Brief Title: Relationship Between Optimal Laryngeal Mask Airway Cuff Volume and Physical Examination of Head and Neck
Acronym: RCVPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Korea University Anam Hospital (Other)
Responsible Party: Principal Investigator, Hye-Won Shin, Director, MD, PhD, Korea University Anam Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: LMA60
Record Dates: First submitted 2015-07-16; First posted 2015-07-20 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Anesthesia
Keywords: Laryngeal mask airway

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Classic laryngeal mask airway (Other): single arm
  Interventions: Device: Classic laryngeal mask airway

INTERVENTIONS:
Device: Classic laryngeal mask airway — 1. measurement of head and neck
     * Ht,Wt,BMI, neck circumference above a thyroid cartilage, mandible circumference( from the lower part of earlobe-mandible angle-mentum-mandible angle to the lower part of earlobe), neck length (mastoid tip~sternal notch), modified mallampati classification under sitting position, thyromental distance.
  2. laryngeal mask airway insertion and measuring cuff pressure by pressure transducer
     * # 4.0 for female, #5.0 for male
     * initial cuff volume(air) : maximum volume recommended by the manufacturer
     * check pressure : if it exceed 60cmH20, we will remove air until 60cmH20
     * remove air until gas leak occured around the cuff under airway pressure 15cmH20, fresh gas flow 6liters/min. Check the volume and pressure just before leakage occured.

SUMMARY:
Overinflation of laryngeal mask airway cuff increase side effect like hoarseness, vocal cord paralysis, sorethroat. The investigators will study correlation between laryngeal mask airway cuff volume and pressure and physical examination of head and neck.

DETAILED DESCRIPTION:
Overinflation of laryngeal mask airway cuff can induce side effects like hoarseness, vocal cord paralysis, sorethroat. Some study revealed that 60cmH2O of intracuff pressure is maximum pressure which is not increase side effect.

The manufacturer recommends that the cuff is inflated with the minimum volume of air required to provide an effective seal(max volume - size 3, 20 ml; size 4, 30 ml; size 5, 40).

The investigators will measure anatomical structure (neck circumference, neck length, thyroid-mental distance, etc.) which can influence cuff volume and pressure and find correlation between cuff volume and physical figure measured.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age 19-65)
* American Society of Anesthesiology Classification I-III

Exclusion Criteria:

* cardiovascular disease, cerebrovascular disease, pulmonary disease
* patient who have operation history for airway
* patient who expected difficult intubation
* patient who have risk of aspiration

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2015-08; Primary Completion 2015-08 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
optimal laryngeal mask airway cuff volume | 20minutes
  ◦The investigators remove air until gas leak occured around the cuff under airway pressure 15cm H20, fresh gas flow 6liters/min. Check the volume and pressure just before leakage occured.

CONTACTS AND LOCATIONS:
Overall Officials: Hye-Won Shin, MD, PhD, Study Director — Department of anesthesiology and pain medicine, Korea University Anam Hospital
Locations (1):
- Korea university anam hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided